Official Title: Perioperative Monitoring of Cardiac Surgery Patients With the Vitalstream Physiological Monitor

NCT05905536

IRB Approved Date: 04/11/24



#### **Informed Consent**

Department/Section of Anesthesiology/Critical Care Medicine

# PERIOPERATIVE MONITORING OF CARDIAC SURGERY PATIENTS WITH THE VITALSTREAM PHYSIOLOGICAL MONITOR

# INFORMED CONSENT FORM TO PARTICIPATE IN RESEARCH

Ashish Khanna, MD, Principal Investigator

#### **SUMMARY**

You are invited to participate in a research study. The purpose of this research study is to evaluate a wrist device called the Vitalstream, a device manufactured by Caretaker Medical, Inc. The Vitalstream is an FDA approved, novel monitoring device that measures vital signs after cardiac surgery in patients in the intensive care unit. We are asking for you to participate in this research study evaluating this device while you are having your surgery as well as during your initial recovery period in the Cardiac Intensive Care Unit (CVICU). We are also asking as a part of this research study to review your medical record to obtain information about your surgery and your treatment in the cardiac intensive care unit.

Participation in this study will involve placing the Vitalstream device on your wrist with a small finger cuff in the holding room on the morning of your surgery. You will also have a small cuff slid on to the same finger that will monitor your oxygen level called a pulse oximeter. This also clips to the Vitalstream device. You will then continue to wear this device throughout your surgery and into the CVICU. Your study participation will end when your surgeon removes some of the monitoring devices you will receive routinely for your surgery. On arrival in the CVICU, and again 3 hours later, research staff will perform what is called a passive leg raise, which is where your leg will be lifted to a 45 degree angle. We will be watching for a change in your vital signs on the Vitalstream device.

The Vitalstream device works just by being attached to your wrist, similar to a smart watch, with a finger cuff that wirelessly measures your blood pressure, heart rate, and your breathing rate. The pulse oximeter will be placed below the cuff mentioned above and will continuously and wirelessly monitor your oxygen level. We are then going to be comparing this information to the information that is in your medical record that was obtained using standard monitoring after heart surgery. You do not have to take any tests or do anything special to be in the study, only allow permission for the study team to place this device and to retrieve your medical information. Your care will not be changed as a result of the use of this device.


Adult Consent Form



All research studies involve some risks. There is the possibility that you may not benefit from your participation in this study and your participation in this study is voluntary. You do not have to allow us to review your medical record if you do not want to. You will not lose any services, benefits, or rights you would normally have if you choose not to participate.

The remainder of this form contains a more complete description of this study. Please read this description carefully. You can ask any questions if you need help deciding whether to join the study. The person in charge of this study is Dr. Ashish Khanna, one of the cardiac intensive care unit medical providers. If you have questions, suggestions, or concerns regarding this study or you want to withdraw from the study, please contact Dr. Khanna at

| If you have any questions, suggestions or | concerns about you | ur rights as a volunteer in this |
|---|---|---|
| research, contact the Institutional Review | Board at | or the Research Subject |
| Advocate at Wake Forest at | | <del></del> |

## **INTRODUCTION**

You are invited to be in a research study. Research studies are designed to gain scientific knowledge that may help other people in the future. You are being asked to take part in this study because you are having cardiac surgery and will be in the CVICU after your surgery. Your participation is voluntary. Please take your time in making your decision as to whether or not you wish to participate. Ask your study doctor or the study staff to explain any words or information contained in this informed consent document that you do not understand. You may also discuss the study with your friends and family.

#### WHY IS THIS STUDY BEING DONE?

The purpose of this research study is to compare the results of the Vitalstream Caretaker device to the standard monitoring devices that are normally used after cardiac surgery. The Caretaker device has been approved by the US Food and Drug Administration (FDA) to be used in this manner.

## HOW MANY PEOPLE WILL TAKE PART IN THE STUDY?

At Wake Forest Baptist Medical Center, we plan to enroll up to 46 patients in this research study.

## WHAT IS INVOLVED IN THE STUDY?

Research staff will approach you prior to your surgery either in the preoperative assessment clinic during your visit to see the anesthesiologist or, if you are a current patient scheduled for surgery, seen in your patient room. This study will be explained in detail. If you wish to participate you will be asked to sign this form.

On the day of your surgery, you will be seen by a member of the research staff in the holding room and have the Vitalstream device placed on your wrist with the pulse oximeter placed on your finger as described earlier. It will then continue to monitor throughout your surgery and into the CVICU for your recovery. After arrival in the CVICU, and again 3 hours after admission, research staff will perform a passive leg raise, when your leg will be lifted 45 degrees


Adult Consent Form



for less than a minute. We will watch for any changes in your vital signs. Your study participation ends when either your surgeon removes your standard of care monitoring devices or at 24 hours, whichever occurs first.

If you agree to participate, as part of the data collection for this study, your electronic medical record will be reviewed and information about your hospital stay will be retrieved. This will include demographic information, information about your surgical procedure and your stay in the cardiac intensive care unit, and medications that you received. The information will also be retrieved from the Caretaker device. All information that is collected will be de-identified and a unique subject identifier used to maintain confidentiality.

## HOW LONG WILL I BE IN THE STUDY?

You will be in the study for the length of time you are admitted to the holding room until the device is removed in the cardiac intensive care unit when your surgeon removes the hemodynamic monitors that are used routinely to track your vital signs. You can stop participating at any time. If you decide to stop participating in the study we encourage you to talk to the investigators or study staff first to learn about any potential health or safety consequences.

## WHAT ARE THE RISKS OF THE STUDY?

Being in this study involves some risk to you. You should discuss the risk of being in this study with the study staff. There is a slight risk of a breach of confidentiality. We will do our best to protect your confidential information. There also may be other risks that we cannot predict. The risk of harm or discomfort that may happen as a result of taking part in this research study is not expected to be more than in daily life or from routine physical or psychological examinations or tests. You should discuss the risk of being in this study with the study staff. Taking part in this research study may involve providing information that you consider confidential or private. Efforts, such as coding research records, keeping research records secure and allowing only authorized people to have access to research records, will be made to keep your information safe.

The Caretaker device is non-invasive and just straps to your wrist like a watch band. The cuff that wraps around your finger uses Velcro to hold itself in place. The pulse oximeter is just a small rubber ring that is placed on your finger below the Vitalstream device that also transfers the information collected to the Caretaker device. Information from this device is downloaded wirelessly to a research computer but is de-identified.

## Reproductive Risks and other Issues to Participating in Research

Pregnant women are excluded from participation in this study. If you are a sexually active woman of childbearing potential and have not been using a reliable method of birth control, a negative urine pregnancy test will be required prior to starting treatment.

#### ARE THERE BENEFITS TO TAKING PART IN THE STUDY?

If you agree to take part in this study, there may or may not be direct benefit to you. We hope the information learned from this study will benefit other people in the future. Our aim is to show that the Caretaker device works just as well as the invasive monitors that are normally used as

Page **3** of **7**Adult Consent Form



standard monitoring for cardiac surgery.

## WHAT OTHER CHOICES ARE THERE?

You do not have to be in this study to receive treatment. You should talk to your doctor about all the choices you have. Instead of being in this study, you have these options: not allowing research personnel to review your medical record to retrieve information about your surgery and recovery.

## WHAT ARE THE COSTS?

Costs for your regular medical care, which are not related to this study, will be your own responsibility. You and/or your insurance company will not be billed for the cost of the use of the Caretaker device.

## WILL YOUR RESEARCH RECORDS BE CONFIDENTIAL?

The results of this research study may be presented at scientific or medical meetings or published in scientific journals. Your identity and/or your personal health information will not be disclosed unless it is authorized by you, required by law, or necessary to protect the safety of yourself or others. There is always some risk that even de-identified information might be re-identified. Participant information may be provided to Federal and other regulatory agencies as required. The Food and Drug Administration (FDA), for example, may inspect research records and learn your identity if this study falls within its jurisdiction.

The results will be provided to the sponsor, the Food and Drug Administration and other federal and regulatory agencies as required.

#### WILL YOU BE PAID FOR PARTICIPATING?

You will receive no payment or other compensation for taking part in this study.

#### WHO IS SPONSORING THIS STUDY?

This study is being sponsored by Caretaker Medical. The sponsor is providing money or other support to Wake Forest University Health Sciences to help conduct this study. The researchers do not, however, hold a direct financial interest in the sponsor or the product being studied.

# WHAT HAPPENS IF YOU EXPERIENCE AN INJURY OR ILLNESS AS A RESULT OF PARTICIPATING IN THIS STUDY?

You do not give up any legal rights as a research participant by signing this consent form. For more information on medical treatment for research related injuries or to report a study related illness, adverse event, or injury you should call Dr. Ashish Khanna at

## WHAT ABOUT MY HEALTH INFORMATION?

In this research study, any information we get from your medical records about your health or behaviors is considered <u>Protected Health Information</u>. The information we will collect for this research study includes information about your hospitalization and the treatments you received during this hospitalization. If this research study involves the diagnosis or treatment of a medical


Adult Consent Form



condition, then Protected Health Information collected from you during this study will be placed in your medical record, and may be used to help treat you, arrange payment for your care, or assist with Medical Center operations. We will make every effort to keep your Protected Health Information private. We will store records of your Protected Health Information in a cabinet in a locked office or on a password-protected computer.

Your personal health information and information that identifies you ("your health information") may be given to others during and after the study. This is for reasons such as to carry out the study, to determine the results of the study, to make sure the study is being done correctly, to provide required reports and to get approval for new products.

Some of the people, agencies and businesses that may receive and use your health information are the research sponsor; representatives of the sponsor assisting with the research (Caretaker Medical); the Institutional Review Board; representatives of Wake Forest University Health Sciences and North Carolina Baptist Hospital; representatives from government agencies such as the Food and Drug Administration (FDA) or the Office of Human Research Protections (OHRP), the Department of Health and Human Services (DHHS) and similar agencies in other countries.

Some of these people, agencies and businesses may further disclose your health information. If disclosed by them, your health information may no longer be covered by federal or state privacy regulations. Your health information may be disclosed if required by law. Your health information may be used to create information that does not directly identify you. This information may be used by other researchers. You will not be directly identified in any publication or presentation that may result from this study unless there are photographs or recorded media which are identifiable.

Monitors, auditors, IRB or other regulatory agencies will be granted direct access to the participant's original medical record for verification of clinical trial procedures or data, without violating confidentiality of the participant and to the extent permitted by other applicable laws.

If required by law or court order, we might also have to share your Protected Health Information with a judge, law enforcement officer, government agencies, or others. If your Protected Health Information is shared with any of these groups it may no longer be protected by federal or state privacy rules.

Any Protected Health Information collected from you for this study that is maintained in the research records will be kept for at least six years after the study is finished. At that time any research information collected specifically for the study will be destroyed.

You can tell Dr. Khanna that you want to take away your permission to use and share your Protected Health Information at any time by sending a letter to this address:





However, if you take away permission to use your Protected Health Information you will not be able to be in the study any longer. We will stop collecting any more information about you, but any information we have already collected can still be used for the purposes of the research study.

By signing this form you give us permission to use your Protected Health Information for this study. If you choose to participate in this study, your medical record at Wake Forest University Baptist Medical Center will indicate that you were enrolled in a clinical trial. Information about the research and any medications or devices you are being given as a participant may also be included in your medical record. This part of the medical record will only be available to people who have authorized access to your medical record. If you are not a patient at this Medical Center, a medical record will be created for you anyway to ensure that this important information is available to doctors in case of an emergency.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this Web site at any time. Laboratory test results and other clinically relevant medical reports created as a result of your participation in the research study may be entered into the computer systems of Wake Forest University Health Sciences and North Carolina Baptist Hospital. These will be kept secure, with access to this information limited to individuals with proper authority, but who may not be directly involved with this research study.

A North Carolina Baptist Hospital (NCBH) medical record will be created for all study participants. Information about your participation in the study will be placed in the NCBH medical record, along with any routine medical test results that were obtained at NCBH as part of this study.

## WHAT ARE MY RIGHTS AS A RESEARCH STUDY PARTICIPANT?

Taking part in this study is voluntary. You may choose not to take part or you may leave the study at any time. Refusing to participate or leaving the study will not result in any penalty or loss of benefits to which you are entitled. If you decide to stop participating in the study we encourage you to talk to the investigators or study staff first to learn about any potential health or safety consequences. The investigators also have the right to stop your participation in the study at any time. This could be because it is in your best medical interest, or your condition worsened. Information that identifies you may be removed from the data or specimens that are collected as part of this study and could be used for future research or shared with others without additional consent. You will be given any new information we become aware of that would affect your willingness to continue to participate in the study.

## WHOM DO I CALL IF I HAVE QUESTIONS OR PROBLEMS?

For questions about the study or in the event of a research-related injury, contact the study investigator, Dr. Ashish Khanna at or by phone at


Adult Consent Form



| The Institutional Review Board (IRB) is a group of people who review the research to p | rotect |
|---|---|
| your rights. If you have a question about your rights as a research participant, or you wo | ould like |
| to discuss problems or concerns, have questions or want to offer input, or you want to of | btain |
| additional information, you should contact the Chairman of the IRB at | or the |
| Research Subject Advocate at | |

You will be given a copy of this signed consent form.

## **SIGNATURES**

I agree to take part in this study. I authorize the use and disclosure of my health information as described in this consent and authorization form. If I have not already received a copy of the Privacy Notice, I may request one or one will be made available to me. I have had a chance to ask questions about being in this study and have those questions answered. By signing this consent and authorization form, I am not releasing or agreeing to release the investigator, the sponsor, the institution or its agents from liability for negligence.

| Subject Name (Printed): | | | |
|-------------------------------------|-------|-------|-------|
| Subject Signature: | Date: | Time: | am pm |
| Person Obtaining Consent (Printed): | | | |
| Person Obtaining Consent: | Date: | Time: | am pn |

 Adult Consent Form